CLINICAL TRIAL: NCT01988610
Title: Effects of Mifepristone on Biomarkers of Metabolic Function and Neuropsychological Performance Among Middle-Aged and Older Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Natalie Rasgon, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26482
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Depression
Keywords: cognition; prediabetes; mood
MeSH Terms: conditions — Depression; Prediabetic State | interventions — Therapeutics; Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Group (Experimental): Open-label trial to assess the effects of Mifepristone on mood and cognition in people with a history of depression.
  Interventions: Drug: 28 days treatment with Mifepristone.

INTERVENTIONS:
Drug: 28 days treatment with Mifepristone.
  Other Names: Korlym; RU486

SUMMARY:
The purpose of this study is to study the effect of cortisol,a stress hormone in the body, on memory and attention in people with a history of depression, but who are not in the midst of a current depressive episode.

Cortisol may affect parts of the brain associated with memory and attention directly. It may also indirectly affect the brain by controlling how much insulin the body makes. Insulin is thought to impact cognition by changing the amount of sugar available in certain parts of the brain.

The investigators are studying this question by giving patients a medication, called Mifepristone, which reduces cortisol's effect on the brain. The investigators will compare results from several groups of people, including differences between men and women, and between those with and without insulin resistance.

DETAILED DESCRIPTION:
The specific aims of this study are threefold:

1. To evaluate the association between glucose utilization and neuropsychological performance on tests of verbal memory and attention among patients with a history of depression, but who are euthymic, at baseline;
2. To evaluate changes in neuropsychological test performance among patients with a history of depression and who have insulin resistance who are treated with open-label mifepristone and,
3. To explore interactions between changes in patients' glucose tolerance profiles and changes in verbal memory and attention. An exploratory aim is to explore the interaction of changes in cortisol awakening response and changes in verbal memory and attention within subjects with and without IGT, as well as the potential mediating effects of gender.

ELIGIBILITY:
Inclusion Criteria:

* Ages 50-70
* History of depression, not currently depressed.

Exclusion Criteria:

* History of type 1 or type 2 diabetes.
* Use of a medication that interacts with Mifepristone.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-10; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Cognition | 3 months
  Neurocognitive testing will assess changes in memory and attention

SECONDARY OUTCOMES:
Hamilton Score | 3 months
  Change in hamilton score as a measure of current mood.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Rasgon, M.D., Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University Psychiatry, 401 Quarry Rd, Stanford, California, United States